CLINICAL TRIAL: NCT01316380
Title: A Phase III, Randomised, Double-blind, Placebo-controlled, Parallel-group Trial to Evaluate Efficacy and Safety of Tiotropium Inhalation Solution Delivered Via Respimat® Inhaler (2.5 ug and 5 ug Once Daily) Compared to Placebo Over 12 Weeks in Mild Persistent Asthma
Brief Title: Efficacy and Safety of 2 Doses of Tiotropium Via Respimat in Adult Patients With Mild Persistent Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.442; 2010-023112-14 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-03-15; First posted 2011-03-16 (Estimated); Results first posted 2013-07-31 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Tiotropium Bromide

ARMS (3):
- tiotropium 5 mcg (Experimental): once daily delivered via Respimat inhaler
  Interventions: Drug: tiotropium 5 mcg
- tiotropium 2.5 mcg (Experimental): once daily delivered via Respimat inhaler
  Interventions: Drug: tiotropium 2.5 mcg
- placebo (Placebo Comparator): once daily delivered via Respimat inhaler
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: placebo — To evaluate efficacy and safety of 2.5 and 5 mcg tiotropium versus placebo delivered via Respimat inhaler
  Arms: placebo
Drug: tiotropium 2.5 mcg — To evaluate efficacy and safety of 2.5 and 5 mcg tiotropium versus placebo delivered via Respimat inhaler
  Arms: tiotropium 2.5 mcg
Drug: tiotropium 5 mcg — To evaluate efficacy and safety of 2.5 and 5 mcg tiotropium versus placebo delivered via Respimat inhaler
  Arms: tiotropium 5 mcg

SUMMARY:
The aim of this trial is to evaluate the efficacy and safety of 2.5 and 5 mcg tiotropium compared to placebo over 12 week treatment period. Tiotropium inhalation solution will be delivered via Respimat inhaler and will be examined on top of maintenance inhaled corticosteroid treatment in patients with mild persistent asthma. Efficacy and safety will be assessed by measuring the effects on lung functions, effects on lung exacerbations, effects on asthma control and numbers of adverse events.

ELIGIBILITY:
Inclusion criteria:

1. All patients must sign and date an Informed Consent Form consistent with International Conference on Harmonisation -Good Clinical Practice (ICH-GCP) guidelines and local legislation prior to participation in the trial (i.e. prior to any trial procedures, including any pre-trial washout of medications and medication restrictions for pulmonary function test at Visit 1).
2. Male or female patients aged 18 years or more at Visit 0 and 75 years or less at Visit 0.

   All patients must have
3. at least a 3 months history of asthma at the time of enrolment into the trial. The initial diagnosis of asthma must have been made before the patient's age of 40;
4. a pre-bronchodilator Forced Expiratory Volume in 1 second (FEV1)= 60% predicted and = 90% of predicted normal at Visit 1. Variation of absolute FEV1 values of Visit 1 (pre-bronchodilator) as compared to Visit 2 (pre-dose) must be within ± 30%.
5. Patient's diagnosis of asthma has to be confirmed at Visit 1 with a bronchodilator reversibility (within 10 minutes pre and 15-30 minutes after 400 µg salbutamol/albuterol) resulting in a FEV1 increase of = 12% and = 200mL. If this is not achieved the reversibility test may be repeated once within two weeks.
6. All patients must be symptomatic despite their current maintenance treatment with low doses of inhaled corticosteroids.
7. All patients must be symptomatic at Visit 1 (screening) and Visit 2 as defined by an Asthma Control Questionnaire (ACQ) mean score of = 1.5.
8. All patients must have been on maintenance treatment with a low, stable dose of inhaled corticosteroids for at least 4 weeks prior to Visit 1.
9. Patients must be never-smokers or ex-smokers who stopped smoking at least one year prior to enrolment and who have a smoking history of less than 10 pack years ((see Appendix 10.3 for calculation).
10. Patients must be able to use the Respimat® inhaler correctly.
11. Patients must be able to perform all trial related procedures including technically acceptable pulmonary function tests and use of the e-Diary/peak flow meter (e-Diary-compliance of at least 80% is required; refer to Section 6.2.1 for instructions).
12. Patients taking a chronic pulmonary medication allowed by the study protocol must be willing to continue this therapy for the entire duration of the study (exception: times of acute disease deterioration).

Exclusion criteria:

1. Patients with a significant disease other than asthma. A significant disease is defined as a disease which, in the opinion of the Investigator, may (i) put the patient at risk because of participation in the trial, or (ii) cause concern regarding the patient's ability to participate in the trial.
2. Patients with a clinically relevant abnormal screening (Visit 1) haematology or blood chemistry if the abnormality defines a significant disease as defined in exclusion criterion number 1.
3. Patients requiring more than 10 puffs of rescue medication (salbutamol/albuterol MDI) per 24 hours on 2 consecutive days during the screening period.
4. Patients with a recent history (i.e. six months or less) of Acute Coronary Syndrome (STEMI, Non-STEMI and Unstable Angina Pectoris).
5. Patients who have been hospitalised for cardiac failure during the past year.
6. Patients with any unstable or life-threatening cardiac arrhythmia or cardiac arrhythmia requiring intervention or a change in drug therapy within the past year.
7. Patients with lung diseases other than asthma (e.g. COPD).
8. Patients with known active tuberculosis.
9. Patients with malignancy for which the patient has undergone resection, radiation therapy or chemotherapy within the last five years. Patients with treated basal cell carcinoma are allowed.
10. Patients who have undergone thoracotomy with pulmonary resection. Patients with a history of thoracotomy for other reasons should be evaluated as per exclusion criterion no.1.
11. Patients with significant alcohol or drug abuse on Investigator's assessment within the past two years.
12. Patients who are currently in a pulmonary rehabilitation program or have completed a pulmonary rehabilitation program in the 6 weeks prior to Visit 1 (screening).
13. Patients with known hypersensitivity to anticholinergic drugs, BAC, EDTA or any other components of the tiotropium inhalation solution.
14. Pregnant or nursing woman, including female patients with positive beta-HCG test at Visit 1.
15. Female patients of child-bearing potential not using highly effective method of birth control As defined in ICH (M3).
16. Patients who have been treated with beta-blocker medication within four weeks prior to Visit 1 and/or during the screening period.Topical cardio-selective beta-blocker eye medications for non-narrow angle glaucoma are allowed.
17. Patients who have been treated with oral or patch beta-adrenergics, systemic, i.e. oral or intravenous corticosteroids, long-acting anticholinergic tiotropium (Spiriva®) within four weeks prior to Visit 1 and/or during the screening period.
18. Patients who have been treated with depot corticosteroids within six months prior to Visit 1 and/or during the screening period.
19. Patients who have ever been treated with anti-IgE antibodies.
20. Patients who have been treated with leukotriene modifiers, systemic anticholinergics, cromolyn sodium or nedocromil sodium and methylxanthines or phosphodiesterase 4 inhibitors within two weeks prior to Visit 1 and/or during the screening period.
21. Patients who have been treated with inhaled long acting beta adrenergics and long acting beta adrenergics combination products within four weeks prior to Visit 0 and/or during the screening period.
22. Patients who have taken an investigational drug within four weeks or six half lives whichever is greater prior to Visit 1.
23. Patients who have been treated with other non-approved and according to international guidelines not recommended, experimental drugs for routine asthma therapy (e.g. TNFalpha blockers, methotrexate, cyclosporin) within four weeks prior to Visit 1 and/or during the screening period (period between Visit 1 and Visit 2).
24. Patients with any asthma exacerbation or any respiratory tract infection in the four weeks prior to Visit 1 and/or during the screening period (period between Visit 1 and Visit 2).
25. Current participation in another trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 465 (Actual)
Dates: Start 2011-03; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (62):
- Argentina (3):
  - 205.442.54002 Boehringer Ingelheim Investigational Site, Capital Federal
  - 205.442.54005 Boehringer Ingelheim Investigational Site, Capital Federal
  - 205.442.54003 Boehringer Ingelheim Investigational Site, San Juan Bautista
- Austria (3):
  - 205.442.43002 Boehringer Ingelheim Investigational Site, Linz
  - 205.442.43003 Boehringer Ingelheim Investigational Site, Schlüsslberg
  - 205.442.43001 Boehringer Ingelheim Investigational Site, Wels
- Croatia (4):
  - 205.442.38502 Boehringer Ingelheim Investigational Site, Rijeka
  - 205.442.38501 Boehringer Ingelheim Investigational Site, Split
  - 205.442.38503 Boehringer Ingelheim Investigational Site, Split
  - 205.442.38504 Boehringer Ingelheim Investigational Site, Zagreb
- Estonia (3):
  - 205.442.37203 Boehringer Ingelheim Investigational Site, Kohtla-Järve
  - 205.442.37201 Boehringer Ingelheim Investigational Site, Rakvere
  - 205.442.37202 Boehringer Ingelheim Investigational Site, Tartu
- Guatemala (5):
  - 205.442.50203 Boehringer Ingelheim Investigational Site, Guatemala City
  - 205.442.50204 Boehringer Ingelheim Investigational Site, Guatemala City
  - 205.442.50201 Boehringer Ingelheim Investigational Site, Nivel Guatemala
  - 205.442.50202 Boehringer Ingelheim Investigational Site, Nivel Guatemala
  - 205.442.50205 Boehringer Ingelheim Investigational Site, Vila Hermosa I
- Hungary (7):
  - 205.442.36007 Boehringer Ingelheim Investigational Site, Budapest
  - 205.442.36003 Boehringer Ingelheim Investigational Site, Cegléd
  - 205.442.36002 Boehringer Ingelheim Investigational Site, Gödöllö
  - 205.442.36004 Boehringer Ingelheim Investigational Site, Komárom
  - 205.442.36006 Boehringer Ingelheim Investigational Site, Pécs
  - 205.442.36001 Boehringer Ingelheim Investigational Site, Szarvas
  - 205.442.36005 Boehringer Ingelheim Investigational Site, Százhalombatta
- India (10):
  - 205.442.91011 Boehringer Ingelheim Investigational Site, Ahmedabad
  - 205.442.91005 Boehringer Ingelheim Investigational Site, Bangalore
  - 205.442.91009 Boehringer Ingelheim Investigational Site, Banglore
  - 205.442.91002 Boehringer Ingelheim Investigational Site, Coimbatore
  - 205.442.91003 Boehringer Ingelheim Investigational Site, Coimbatore
  - 205.442.91004 Boehringer Ingelheim Investigational Site, Coimbatore
  - 205.442.91008 Boehringer Ingelheim Investigational Site, Hyderabad
  - 205.442.91007 Boehringer Ingelheim Investigational Site, Jaipur
  - 205.442.91001 Boehringer Ingelheim Investigational Site, Nagpur
  - 205.442.91006 Boehringer Ingelheim Investigational Site, Pune
- Italy (4):
  - 205.442.39007 Boehringer Ingelheim Investigational Site, Acquaviva Delle Fonti (BA)
  - 205.442.39006 Boehringer Ingelheim Investigational Site, Cagliari
  - 205.442.39003 Boehringer Ingelheim Investigational Site, Chieti
  - 205.442.39001 Boehringer Ingelheim Investigational Site, Pisa
- Latvia (4):
  - 205.442.37101 Boehringer Ingelheim Investigational Site, Baldone
  - 205.442.37103 Boehringer Ingelheim Investigational Site, Daugavpils
  - 205.442.37104 Boehringer Ingelheim Investigational Site, Daugavpils
  - 205.442.37102 Boehringer Ingelheim Investigational Site, Talsi
- Poland (5):
  - 205.442.48003 Boehringer Ingelheim Investigational Site, Giżycko
  - 205.442.48002 Boehringer Ingelheim Investigational Site, Gorzów Wielkopolski
  - 205.442.48005 Boehringer Ingelheim Investigational Site, Krakow
  - 205.442.48004 Boehringer Ingelheim Investigational Site, Ostrow Wielkopolska
  - 205.442.48001 Boehringer Ingelheim Investigational Site, Poznan
- Slovakia (8):
  - 205.442.42105 Boehringer Ingelheim Investigational Site, Bardejov
  - 205.442.42107 Boehringer Ingelheim Investigational Site, Humenné
  - 205.442.42104 Boehringer Ingelheim Investigational Site, Košice
  - 205.442.42102 Boehringer Ingelheim Investigational Site, Nitra
  - 205.442.42101 Boehringer Ingelheim Investigational Site, Nové Zámky
  - 205.442.42108 Boehringer Ingelheim Investigational Site, Poprad
  - 205.442.42106 Boehringer Ingelheim Investigational Site, Spišská Nová Ves
  - 205.442.42103 Boehringer Ingelheim Investigational Site, Topoľčany
- South Korea (6):
  - 205.442.82006 Boehringer Ingelheim Investigational Site, Cheongju-si
  - 205.442.82002 Boehringer Ingelheim Investigational Site, Gangwon-do
  - 205.442.82001 Boehringer Ingelheim Investigational Site, Seoul
  - 205.442.82003 Boehringer Ingelheim Investigational Site, Seoul
  - 205.442.82004 Boehringer Ingelheim Investigational Site, Seoul
  - 205.442.82005 Boehringer Ingelheim Investigational Site, Seoul

REFERENCES:
- [Derived] Oba Y, Anwer S, Maduke T, Patel T, Dias S. Effectiveness and tolerability of dual and triple combination inhaler therapies compared with each other and varying doses of inhaled corticosteroids in adolescents and adults with asthma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD013799. doi: 10.1002/14651858.CD013799.pub2. PMID 36472162
- [Derived] Halpin DMG, Hamelmann EH, Frith PA, Moroni-Zentgraf PM, van Hecke B, Unseld A, Kerstjens HAM, Szefler SJ. Comparative Responses in Lung Function Measurements with Tiotropium in Adolescents and Adults, and Across Asthma Severities: A Post Hoc Analysis. Pulm Ther. 2020 Jun;6(1):131-140. doi: 10.1007/s41030-020-00113-w. Epub 2020 Mar 16. PMID 32180164
- [Derived] Halpin DMG, Meltzer EO, Pisternick-Ruf W, Moroni-Zentgraf P, Engel M, Zaremba-Pechmann L, Casale T, FitzGerald JM. Peak expiratory flow as an endpoint for clinical trials in asthma: a comparison with FEV1. Respir Res. 2019 Jul 18;20(1):159. doi: 10.1186/s12931-019-1119-6. PMID 31319851
- [Derived] Paggiaro P, Halpin DM, Buhl R, Engel M, Zubek VB, Blahova Z, Moroni-Zentgraf P, Pizzichini E. The Effect of Tiotropium in Symptomatic Asthma Despite Low- to Medium-Dose Inhaled Corticosteroids: A Randomized Controlled Trial. J Allergy Clin Immunol Pract. 2016 Jan-Feb;4(1):104-13.e2. doi: 10.1016/j.jaip.2015.08.017. Epub 2015 Nov 7. PMID 26563670

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Patients treated with matching placebo
- Tio R2.5: Patients treated with tiotropium inhalation solution 2.5 microgram qd
- Tio R5: Patients treated with tiotropium inhalation solution 5 microgram qd
Period: Overall Study
Arm/Group | Placebo | Tio R2.5 | Tio R5
Started | 156 | 154 | 155
Completed | 154 | 149 | 152
Not Completed | 2 | 5 | 3
Not completed — Adverse Event | 0 | 2 | 1
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2 | 0
Not completed — Other | 0 | 1 | 1
Not completed — Not treated | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tio R2.5 | Tio R5 | Total
Number analyzed (Participants) | 155 | 154 | 155 | 464
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.8 (12.1) | 43.8 (14.0) | 41.9 (13.0) | 42.9 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 82 | 96 | 281
  Male | 52 | 72 | 59 | 183

OUTCOME MEASURES:

1. Primary Outcome: Peak Forced Expiratory Volume in 1 Second (FEV1) Response Within 3 Hours Post Dosing (0-3h) After a Treatment Period of 12 Weeks.
Description: Peak FEV1 0-3h response was defined as the difference between the maximum FEV1 measured within the first 3 hours post dosing after a treatment period of 12 weeks and the FEV1 baseline measurement (10 minutes before the first dose of trial medication). Mixed Model Repeated Measure (MMRM) results. Means are adjusted for treatment, pooled centre, visit, baseline, treatment*visit and baseline*visit.
Time Frame: Baseline and 12 weeks
Population: All patients from Full Analysis Set (FAS) FAS is defined as all patients in the treated set who received at least one dose of randomized trial medication.
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Tio R2.5 | Tio R5
Number analyzed (Participants) | 154 | 151 | 152
Liter | 0.134 (0.026) | 0.293 (0.026) | 0.262 (0.026)
Statistical Analysis 1: Comparison: Placebo vs Tio R5; Test type: Superiority or Other; p = 0.0005, Mixed Models Analysis — Step-wise testing for the two treatment groups for the primary endpoint, confirmatory only if previous hypotheses had been successful, significance level of alpha=0.025 (one-sided) for primary endpoint; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Mean Difference (Final Values) = 0.128, 95% CI [0.057 to 0.199], Standard Error of Mean 0.036 — Tio R5 - Placebo. Means are adjusted for treatment, pooled centre, visit, baseline, treatment*visit and baseline*visit
Statistical Analysis 2: Comparison: Placebo vs Tio R2.5; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Step-wise testing for the two treatment groups for the primary endpoint, confirmatory only if previous hypotheses had been successful, significance level of alpha=0.025 (one-sided) for the primary endpoint; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Mean Difference (Final Values) = 0.159, 95% CI [0.088 to 0.230], Standard Error of Mean 0.036 — Tio R2.5 - Placebo. Means are adjusted for treatment, pooled centre, visit, baseline, treatment*visit and baseline*visit

2. Secondary Outcome: Trough FEV1 Response Determined After a Treatment Period of 12 Weeks.
Description: The trough FEV1 is defined as the pre-dose FEV1 measured 10 minutes before the last administration of randomised treatment. Trough FEV1 response was defined as the difference between the trough FEV1 measured after a treatment period of 12 weeks and the trough FEV1 baseline measurement. MMRM results. Means are adjusted for treatment, pooled centre, visit, baseline, treatment*visit and baseline*visit.
Time Frame: Baseline and 12 weeks
Population: All patients from FAS.
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Tio R2.5 | Tio R5
Number analyzed (Participants) | 154 | 151 | 152
Liter | 0.015 (0.026) | 0.125 (0.026) | 0.137 (0.027)
Statistical Analysis 1: Comparison: Placebo vs Tio R5; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis — p-values serve an exploratory function only; REML-based repeated measures approach (MMRM); Mean Difference (Final Values) = 0.122, 95% CI [0.049 to 0.194], Standard Error of Mean 0.037 — Tio R5 - Placebo. Means are adjusted for treatment, pooled centre, visit, baseline, treatment*visit and baseline*visit
Statistical Analysis 2: Comparison: Placebo vs Tio R2.5; Test type: Superiority or Other; p = 0.0028, Mixed Models Analysis — p-values serve an exploratory function only; REML-based repeated measures approach (MMRM); Mean Difference (Final Values) = 0.110, 95% CI [0.038 to 0.182], Standard Error of Mean 0.037 — [estimate comment as in outcome 1, analysis 2]

3. Secondary Outcome: Peak (Within 3 Hours Post-dosing) Forced Vital Capacity (FVC) Response at the End of the 12-week Treatment Period.
Description: Peak FVC 0-3h response was defined as the difference between the maximum FVC measured within the first 3 hours post dosing after a treatment period of 12 weeks and the FVC baseline measurement (10 minutes before the first dose of trial medication). Mixed Model Repeated Measure (MMRM) results. Means are adjusted for treatment, pooled centre, visit, baseline, treatment*visit and baseline*visit.
Time Frame: Baseline and 12 weeks
Population: All patients from FAS.
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Tio R2.5 | Tio R5
Number analyzed (Participants) | 154 | 151 | 152
Liter | 0.126 (0.030) | 0.231 (0.030) | 0.183 (0.03)
Statistical Analysis 1: Comparison: Placebo vs Tio R5; Test type: Superiority or Other; p = 0.1714, Mixed Models Analysis — p-values serve an exploratory function only; REML-based repeated measures approach (MMRM); Mean Difference (Final Values) = 0.057, 95% CI [-0.025 to 0.140], Standard Error of Mean 0.042 — Tio R5 - Placebo. Means are adjusted for treatment, pooled centre, visit, baseline, treatment*visit and baseline*visit
Statistical Analysis 2: Comparison: Placebo vs Tio R2.5; Test type: Superiority or Other; p = 0.0119, Mixed Models Analysis — p-values serve an exploratory function only; REML-based repeated measures approach (MMRM); Mean Difference (Final Values) = 0.106, 95% CI [0.023 to 0.188], Standard Error of Mean 0.042 — [estimate comment as in outcome 1, analysis 2]

4. Secondary Outcome: FEV1 Area Under the Curve (AUC0-3h) Response at the End of the 12-week Treatment Period.
Description: The AUC0-3h was calculated as area under the curve from zero to 3 hours using the trapezoidal rule divided by the observation time (3 hours) to report in litres. The trough value was assigned to zero time. Response was defined as change from baseline in FEV1 AUC0-3h after a treatment period of 12 weeks. MMRM results. Means are adjusted for treatment, pooled centre, visit, baseline, treatment*visit baseline*visit.
Time Frame: Baseline and 12 weeks
Population: All patients from FAS.
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Tio R2.5 | Tio R5
Number analyzed (Participants) | 154 | 151 | 152
Liter | 0.048 (0.024) | 0.198 (0.024) | 0.174 (0.025)
Statistical Analysis 1: Comparison: Placebo vs Tio R5; Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis — p-values serve an exploratory function only; REML-based repeated measures approach (MMRM); Mean Difference (Final Values) = 0.125, 95% CI [0.058 to 0.192], Standard Error of Mean 0.034 — Tio R5 - Placebo. Means are adjusted for treatment, pooled centre, visit, baseline, treatment*visit and baseline*visit
Statistical Analysis 2: Comparison: Placebo vs Tio R2.5; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — p-values serve an exploratory function only; REML-based repeated measures approach (MMRM); Mean Difference (Final Values) = 0.149, 95% CI [0.082 to 0.216], Standard Error of Mean 0.034 — [estimate comment as in outcome 1, analysis 2]

5. Secondary Outcome: FVC (AUC0-3h) Response at the End of the 12-week Treatment Period.
Description: The AUC0-3h was calculated as area under the curve from zero to 3 hours using the trapezoidal rule divided by the observation time (3 hours) to report in litres. The trough value was assigned to zero time. Response was defined as change from baseline in FVC AUC0-3h after a treatment period of 12 weeks. MMRM results. Means are adjusted for treatment, pooled centre, visit, baseline, treatment*visit baseline*visit.
Time Frame: Baseline and 12 weeks
Population: All patients from FAS.
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Tio R2.5 | Tio R5
Number analyzed (Participants) | 154 | 151 | 152
Liter | -0.000 (0.028) | 0.101 (0.028) | 0.061 (0.028)
Statistical Analysis 1: Comparison: Placebo vs Tio R5; Test type: Superiority or Other; p = 0.1182, Mixed Models Analysis — p-values serve an exploratory function only; REML-based repeated measures approach (MMRM); Mean Difference (Final Values) = 0.061, 95% CI [-0.016 to 0.138], Standard Error of Mean 0.039 — Tio R5 - Placebo. Means are adjusted for treatment, pooled centre, visit, baseline, treatment*visit and baseline*visit
Statistical Analysis 2: Comparison: Placebo vs Tio R2.5; Test type: Superiority or Other; p = 0.0102, Mixed Models Analysis — p-values serve an exploratory function only; REML-based repeated measures approach (MMRM); Mean Difference (Final Values) = 0.101, 95% CI [0.024 to 0.178], Standard Error of Mean 0.039 — [estimate comment as in outcome 1, analysis 2]

6. Secondary Outcome: Asthma Control Questionnaire (ACQ) Responder After 12 Weeks of Treatment
Description: For the ACQ, the total score was calculated as the mean of the responses to 6 self administered questions and one question which was completed by clinical staff based upon pre-bronchodilator FEV1. The score ranges from 0 (no impairment) to 6 (maximum impairment). Response was categorised as: responder (change from baseline <= -0.5), no change (-0.5 <change from baseline < 0.5) and worsening (change from baseline >= 0.5).
Time Frame: 12 weeks
Population: All patients from FAS.
Measure: Number; unit: Number of patients
Arm/Group | Placebo | Tio R2.5 | Tio R5
Number analyzed (Participants) | 154 | 149 | 152
Number of patients
  Responder | 91 | 91 | 90
  No change | 61 | 48 | 57
  Worsening | 2 | 10 | 5

7. Secondary Outcome: Time to First Severe Asthma Exacerbation During the 12-week Treatment.
Description: Severe asthma exacerbations are defined as all asthma exacerbations that required treatment with systemic (including oral) corticosteroids for at least 3 days.
Time Frame: 12 weeks
Population: All patients from FAS.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Placebo | Tio R2.5 | Tio R5
Number analyzed (Participants) | 155 | 154 | 155
Days | NA [NA to NA] — Since only 4 of the 155 patients in the placebo group, 6 of the 154 patients in the Tio R2.5 group and 1 of the 155 patients in the Tio R5 group had severe exacerbations, the median times were not calculable (nc). | NA [NA to NA] — Since only 4 of the 155 patients in the placebo group, 6 of the 154 patients in the Tio R2.5 group and 1 of the 155 patients in the Tio R5 group had severe exacerbations, the median times were not calculable (nc). | NA [NA to NA] — Since only 4 of the 155 patients in the placebo group, 6 of the 154 patients in the Tio R2.5 group and 1 of the 155 patients in the Tio R5 group had severe exacerbations, the median times were not calculable (nc).
Statistical Analysis 1: Comparison: Placebo vs Tio R5; Since the percent patients with event is less than 50% the median is not calculable, but Hazard Ratio is still estimable from the Cox model; Test type: Superiority or Other; p = 0.2155, Regression, Cox — Significance level of alpha=0.05 (two-sided). P-values serve an exploratory function only; Parameter estimates of Cox proportional hazard model regarding. Only treatment was fitted as an effect in the model; Hazard Ratio (HR) = 0.25, 95% CI [0.03 to 2.24] — If HR is below 1 then favours tiotropium
Statistical Analysis 2: Comparison: Placebo vs Tio R2.5; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.5071, Regression, Cox — Significance level of alpha=0.05 (two-sided). P-values serve an exploratory function only; Parameter estimates of Cox proportional hazard model regarding. Only treatment was fitted as an effect in the model; Hazard Ratio (HR) = 1.53, 95% CI [0.43 to 5.44] — If HR is below 1 then favours tiotropium

8. Secondary Outcome: Time to First Asthma Exacerbation During the 12-week Treatment.
Description: An asthma exacerbation was defined as an episode of progressive increase in 1 or more asthma symptom that were outside the patient's usual range of day-to-day asthma symptoms and lasted for at least 2 consecutive days or as a decrease in a patient's best morning PEF of 30% or more from a patient's mean morning PEF for at least 2 consecutive days that may or may not have been accompanied by symptoms.
Time Frame: 12 weeks
Population: All patients from FAS.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Placebo | Tio R2.5 | Tio R5
Number analyzed (Participants) | 155 | 154 | 155
Days | NA [87.0 to NA] — Since 22 of the 155 in the placebo group, 21 of the 154 patients in the Tio R2.5 group and 13 of the 155 patients in the Tio R5 group reported at least one asthma exacerbation, the median times were not calculable (nc). | NA [NA to NA] — Since 22 of the 155 in the placebo group, 21 of the 154 patients in the Tio R2.5 group and 13 of the 155 patients in the Tio R5 group reported at least one asthma exacerbation, the median times were not calculable (nc). | NA [NA to NA] — Since 22 of the 155 in the placebo group, 21 of the 154 patients in the Tio R2.5 group and 13 of the 155 patients in the Tio R5 group reported at least one asthma exacerbation, the median times were not calculable (nc).
Statistical Analysis 1: Comparison: Placebo vs Tio R5; Since only 22 of the 155 patients in the placebo group, 21 of the 154 patients in the Tio R2.5 group and 13 of the 155 patients in the Tio R5 group had asthma exacerbations, the median times were not calculable (nc); Test type: Superiority or Other; p = 0.1217, Regression, Cox — Significance level of alpha=0.05 (two-sided). P-values serve an exploratory function only; Parameter estimates of Cox proportional hazard model regarding. Only treatment was fitted as an effect in the model; Hazard Ratio (HR) = 0.58, 95% CI [0.29 to 1.16] — If HR is below 1 then favours tiotropium
Statistical Analysis 2: Comparison: Placebo vs Tio R2.5; Since only 22 of the 155 patients in the placebo group, 21 of the 154 patients in the Tio R2.5 group and 13 of the 155 patients in the Tio R5 group had asthma exacerbations, the median times were not calculable (nc). The Hazard Ratio is still estimable from the Cox model; Test type: Superiority or Other; p = 0.8974, Regression, Cox — Significance level of alpha=0.05 (two-sided). P-values serve an exploratory function only; Parameter estimates of Cox proportional hazard model regarding. Only treatment was fitted as an effect in the model; Hazard Ratio (HR) = 0.96, 95% CI [0.53 to 1.75] — If HR is below 1 then favours tiotropium

9. Secondary Outcome: Use of Rescue Medication During 24h Period
Description: Use of PRN (pro re nata, or as necessary) salbutamol/albuterol rescue medication (puffs during 24 h period), determined as a weekly mean response from baseline for each week during the treatment period as well as for the last 7 days before treatment stop/Visit 5.
  The mean was adjusted for treatment, centre, week, baseline, treatment*week and baseline*week.
Time Frame: Baseline and 12 weeks
Population: All patients from FAS.
Measure: Mean (Standard Error); unit: puffs of rescue medication
Arm/Group | Placebo | Tio R2.5 | Tio R5
Number analyzed (Participants) | 153 | 150 | 152
puffs of rescue medication | -0.815 (0.093) | -0.594 (0.093) | -0.848 (0.093)
Statistical Analysis 1: Comparison: Placebo vs Tio R2.5; Restricted maximum likelihood (REML)- based repeated measures model was used; Test type: Superiority or Other; p = 0.0872, Mixed Models Analysis — p-values serve an exploratory function only; Mean Difference (Net) = 0.222, 95% CI 2-sided [-0.032 to 0.476], Standard Error of Mean 0.129 — Tio R2.5 - Placebo. Means are adjusted for treatment, centre, week, baseline, treatment*week and baseline*week
Statistical Analysis 2: Comparison: Placebo vs Tio R5; Restricted maximum likelihood (REML)- based repeated measures model was used; Test type: Superiority or Other; p = 0.7995, Mixed Models Analysis — p-values serve an exploratory function only; Mean Difference (Net) = -0.033, 95% CI 2-sided [-0.287 to 0.221], Standard Error of Mean 0.129 — Tio R5 - Placebo. Means are adjusted for treatment, centre, week, baseline, treatment*week and baseline*week

10. Secondary Outcome: Use of Rescue Medication During Daytime
Description: Use of PRN (pro re nata, or as necessary) salbutamol/albuterol rescue medication (puffs during daytime), determined as a weekly mean response from baseline for each week during the treatment period as well as for the last 7 days before treatment stop/Visit 5.
  The mean was adjusted for treatment, centre, week, baseline, treatment*week and baseline*week.
Time Frame: Baseline and 12 weeks
Population: All patients from FAS.
Measure: Mean (Standard Error); unit: puffs of rescue medication
Arm/Group | Placebo | Tio R2.5 | Tio R5
Number analyzed (Participants) | 153 | 149 | 152
puffs of rescue medication | -0.428 (0.055) | -0.331 (0.055) | -0.436 (0.055)
Statistical Analysis 1: Comparison: Placebo vs Tio R2.5; Restricted maximum likelihood (REML)- based repeated measures model was used. Means are adjusted for treatment, centre, week, baseline, treatment*week and baseline*week; Test type: Superiority or Other; p = 0.2038, Mixed Models Analysis — p-values serve an exploratory function only; Mean Difference (Net) = 0.097, 95% CI 2-sided [-0.053 to 0.247], Standard Error of Mean 0.076 — Tio R2.5 - Placebo. Means are adjusted for treatment, centre, week, baseline, treatment*week and baseline*week
Statistical Analysis 2: Comparison: Placebo vs Tio R5; Restricted maximum likelihood (REML)- based repeated measures model was used; Test type: Superiority or Other; p = 0.9104, Mixed Models Analysis — p-values serve an exploratory function only; Mean Difference (Net) = -0.009, 95% CI 2-sided [-0.158 to 0.141], Standard Error of Mean 0.076 — Tio R5 - Placebo. Means are adjusted for treatment, centre, week, baseline, treatment*week and baseline*week

11. Secondary Outcome: Use of Rescue Medication During Nighttime
Description: Use of PRN (pro re nata, or as necessary) salbutamol/albuterol rescue medication (puffs during nighttime), determined as a weekly mean response from baseline for each week during the treatment period as well as for the last 7 days before treatment stop/Visit 5.
  The mean was adjusted for treatment, centre, week, baseline, treatment*week and baseline*week.
Time Frame: Baseline and 12 weeks
Population: All patients from FAS.
Measure: Mean (Standard Error); unit: puffs of rescue medication
Arm/Group | Placebo | Tio R2.5 | Tio R5
Number analyzed (Participants) | 152 | 150 | 152
puffs of rescue medication | -0.376 (0.049) | -0.245 (0.049) | -0.386 (0.049)
Statistical Analysis 1: Comparison: Placebo vs Tio R2.5; Restricted maximum likelihood (REML)- based repeated measures model was used; Test type: Superiority or Other; p = 0.0559, Mixed Models Analysis — p-values serve an exploratory function only; Mean Difference (Net) = 0.131, 95% CI 2-sided [-0.003 to 0.265], Standard Error of Mean 0.068 — Tio R2.5 - Placebo. Means are adjusted for treatment, centre, week, baseline, treatment*week and baseline*week
Statistical Analysis 2: Comparison: Placebo vs Tio R5; Restricted maximum likelihood (REML)- based repeated measures model was used; Test type: Superiority or Other; p = 0.8795, Mixed Models Analysis — p-values serve an exploratory function only; Mean Difference (Net) = -0.010, 95% CI 2-sided [-0.144 to 0.123], Standard Error of Mean 0.068 — Tio R5 - Placebo. Means are adjusted for treatment, centre, week, baseline, treatment*week and baseline*week

ADVERSE EVENTS:
Time Frame: 12 weeks
Groups:
- Placebo; Tio R2.5; Tio R5: Enter description here, if needed
Arm/Group | Placebo | Tio R2.5 | Tio R5
Serious Adverse Events (participants affected / at risk) | 1/155 | 0/154 | 1/155
Other Adverse Events (participants affected / at risk) | 25/155 | 30/154 | 21/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=155) | Tio R2.5 (N=154) | Tio R5 (N=155)
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=155) | Tio R2.5 (N=154) | Tio R5 (N=155)
Asthma (Respiratory, thoracic and mediastinal disorders) | 19 | 24 | 17
Peak expiratory flow rate decreased (Investigations) | 6 | 9 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.